CLINICAL TRIAL: NCT05426746
Title: A First-in-human, Phase 1, Randomised, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of Intravenously Infused ALT-100 in Healthy Volunteers
Brief Title: First-In-Human Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ALT-100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aqualung Therapeutics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-100-001
Record Dates: First submitted 2022-06-13; First posted 2022-06-22 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: ARDS, Human
Keywords: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: First in human, randomized, double-blind, placebo-controlled, multi-cohort healthy volunteer trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Site, Clinical Research Organization and Sponsor personnel are are blinded except for unblinded pharmacist staff, unblinded Project Manager, unblinded Monitor and unblinded statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALT-100 (Experimental): one of 4 ascending dose levels of ALT-100 administered as a single intravenous infusion with a staggered dose for sentinels followed by the rest of the cohort.
  cohort 1: 0.1 mg/kg cohort 2: 0.4 mg/kg cohort 3: 1.0 mg/kg cohort 4: 4.0 mg/kg
  Interventions: Drug: ALT-100
- Saline (Placebo Comparator): normal sterile saline (0.9% sodium chloride) administered as a single intravenous infusion at a constant infusion rate in a total volume and appearance matched to the active comparator, with a staggered dose for sentinels followed by the rest of the cohort
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: ALT-100 — intravenous infusion of drug substance diluted in 0.9% normal sterile saline
  Arms: ALT-100
Other: Normal Saline — intravenous infusion of placebo (0.9% normal sterile saline)
  Arms: Saline

SUMMARY:
ALT-100 is a monoclonal antibody developed by Aqualung Therapeutics Corp. as a treatment for Acute Respiratory Distress Syndrome (ARDS). ARDS can occur as a serious complication in patients with respiratory infections such as COVID-19 and Influenza or have acquired trauma to their lungs. 32 healthy male or female participants between the ages of 18 and 55 years will be enrolled into 4 cohorts of single ascending doses. The doses being investigated are 0.1mg/kg, 0.4mg/kg, 1mg/kg and 4mg/kg administered by intravenous infusion. Participants will be screened within 28 days of study treatment, be admitted to the clinical research unit for 3 nights and attend 7 outpatient visits on study days 8, 15, 22, 29, 60, 90 and 120 respectively. This study will collect data to evaluate safety and tolerability, Pharmacokinetics of ALT-100, Pharmacodynamics of ALT-100 and determine if Anti-drug Antibodies are produced in the participants.

DETAILED DESCRIPTION:
Inflammation is a key feature in the pathogenesis of sepsis and ARDS. The investigational product (IP), ALT-100, is a humanised murine mAb that binds specifically to eNAMPT, a novel therapeutic target for ARDS and ARDS associated ventilator-induced lung injury (VILI). ALT-100 is proposed for development as a potential treatment for patients with ARDS and VILI.

This is a first-in-human (FIH), Phase 1, randomised, double-blind, placebo-controlled study to investigate the safety, tolerability, and PK profile of single ascending doses of IV infused ALT-100 administered in healthy participants. The PD effects of ALT-100 will also be explored.

The Single ascending dose escalation study will be conducted in approximately 32 evaluable participants who will be sequentially enrolled and randomised in a 3:1 ratio (active: placebo) to one of 4 planned single ascending dose (SAD) cohorts:

* Cohort 1: 0.1 (mg/kg) ALT-100 (6 participants)/ Placebo (2 participants)
* Cohort 2: 0.4 (mg/kg) ALT-100 (6 participants)/ Placebo (2 participants)
* Cohort 3: 1.0 (mg/kg) ALT-100 (6 participants)/ Placebo (2 participants)
* Cohort 4: 4.0 (mg/kg) ALT-100 (6 participants)/ Placebo (2 participants)

A sentinel dosing strategy will be utilised for the first 2 participants (n=1 active; n=1 placebo) in each dosing cohort. Sentinel participants will receive study drug at least 14 days before the remainder of participants in the cohort. In the absence of clinically significant safety signals in sentinel participants over the 14-day post-treatment observation period (up to and including the Day 15 visit, as determined by the Investigator, in consultation with the local medical monitor (MM) and Sponsor if required), the remainder of participants in the cohort may proceed to be admitted, randomised and dosed, at the Investigator's discretion, with a sufficient minimum interval between all subsequent participants to allow monitoring of any acute post-dose safety events.

Screening (Day -29 to Day -2) and Admission (Day -1): Screening for the study will occur within 28 days prior to enrolment and admission on Day -1 to the clinical research unit (CRU). Informed consent must be documented before any study-specific procedure, including for screening, is performed. Consenting participants who meet all the eligibility criteria at screening will be enrolled upon confirmation of their eligibility at the time of admission to the CRU on Day -1. Participants will be randomised on the morning of Day 1 to receive ALT-100 or placebo by IV infusion. All participants will undergo baseline assessments prior to administration of study treatment on Day 1. Screening and baseline assessments are outlined in the Schedule of Assessments (SOA).

Treatment (Day 1): Randomised study participants will be administered a single IV infusion of study drug per their assigned treatment on Day 1. Following study drug administration on Day 1, all participants will remain confined at the CRU and will undergo safety, PK, PD and other assessments, per the Schedule of Assessments.

In the absence of clinically significant safety signals, and at the Investigator's discretion, participants will be discharged from the CRU on Day 3 following completion of all specified assessments.

Participants will return to the CRU on an outpatient basis on Day 8 (±1 day), Day 15 (±1 day), Day 22 (±2 days), Day 29 (±3 days), Day 60 (±7 days), Day 90 (±7 days) and at Day 120 (±7 days) for safety and other assessments.

Additional unscheduled visits may occur at the Investigator's discretion, i.e., if considered necessary for clinical safety reasons

The Day 120 visit will constitute the end of study participation. A participant will be considered to have completed the study following completion of all assessments at the Day 120 visit.

Early termination: In the case of premature discontinuation from the study, participants will return to the CRU and complete an early termination (ET) visit. For participants who withdraw prior to Day 29, assessments conducted at the ET visit will be as described for the onsite visit on Day 29 (±3 days). For participants who withdraw after Day 29, assessments conducted at the ET visit will be as described for the onsite visit on Day 120 (±7 days). All participants who withdraw from the study early will be followed up for at least 28 days (±3 days) after administration of the study drug unless participant consent is withdrawn.

Safety Oversight :The study will be subject to oversight by an SMC comprised of the Principal Investigator (PI), local MM, and Sponsor medical representative as core members.

The SMC will convene for each SAD dosing cohort to determine if dose escalation may proceed based on review of cumulative data. This will include, at a minimum, review of 28 days of post-treatment safety data (i.e., safety data up to and including the Day 29 visit) and all available PK data from the ongoing cohort as well as the accumulated data from all previous cohorts (where applicable). Where a participant is withdrawn from the study before Day 29, all available safety and PK data up to the time of withdrawal will be reviewed by the SMC. Data from participants receiving placebo and active treatment will be considered in the dose escalation discussion. The dose escalation decision will be based upon the nature, severity and frequency of any safety and/or tolerability observations, and the safety data will include any AEs or SAEs, ECG and vital sign and safety laboratory changes, and physical findings.

Dose escalation: The SMC may recommend escalation to the next dose, escalation to an intermediate dose (a dose lower than the next planned dose), continuation or delay in dosing, repetition or expansion of a cohort, de-escalation to a lower dose, or termination of the study. The SMC may also recommend additional SAD dose cohorts, or they may pause the study to conduct an expert review and to determine next steps. Dose escalation decisions may be delayed to allow collection of additional data if indicated (e.g., safety and/ or PK data).

No intra-cohort dose escalation is permitted.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 55 years of age, inclusive.
2. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, safety laboratory tests and cardiac monitoring at screening and admission. Potential participants with a history of childhood asthma (resolved), depression (non-hospitalised, but potentially medicated in the past) and migraine may be considered for study participation. A potential participant with a clinical abnormality or laboratory parameters outside the normal reference range for the population being studied may be rescreened once, at the Investigator's discretion, and may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. The Investigator may discuss with the local MM and Sponsor medical representative as required.
3. Normal vital signs after greater than or equal to 5 minutes resting in a supine or semi-supine position:

   1. greater than 90 mmHg and less than 160 mmHg systolic blood pressure (SBP)
   2. greater than 50 mmHg and less than 95 mmHg diastolic blood pressure (DBP)
   3. greater than 45 bpm and less than 100 bpm heart rate (HR)
   4. Body temperature greater than or equal to 35.5°C to less than or equal to 37.7°C
4. Standard 12-lead ECG parameters after greater than or equal to 5 minutes resting in a supine or semi-supine position with PR greater than 120 msec and less than 220 msec, QRS less than 120 msec, QT Interval with Fridericia's Correction (QTcF) less than or equal to450 msec for males and less than or equal to 470 msec for females, and otherwise normal ECG.
5. Normal creatinine clearance values (>60 mL/min) at screening (calculated from serum creatinine by a predicting equation using Cockcroft-Gault formula), normal serum creatinine value as defined by the local reference laboratory, normal urine microscopy and no significant proteinuria on dipstick testing.
6. Body weight greater than or equal to 50 kg and BMI in the range 18 kg/m2 - 32 kg/m2 (inclusive).
7. Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or use highly effective contraceptive method (oral contraceptive pills [OCPs], long-acting implantable hormones, injectable hormones, a vaginal ring or an intrauterine device [IUD]) from screening until study completion, including the follow up period for at least 30 days after the last dose of study drug, or be post-menopausal for greater than or equal to 12 months. Post-menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels (greater than or equal to 40 IU/L) at screening for amenorrheic female participants. Female participants who's only partner has had a vasectomy, and female participants who are abstinent from heterosexual intercourse as part of their usual lifestyle will also be eligible for participation.
8. Women of child-bearing potential (WOCBP) must have a negative pregnancy test at screening and admission and be willing to have additional pregnancy tests as required throughout the study.
9. Males must be surgically sterile (greater than 30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a WOCBP, the male participant and his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) and/ or using an acceptable, highly effective contraceptive method from screening until study completion, including the follow up period, for at least 90 days after the last dose of study drug. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner (WOCBP) that includes: OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring or an IUD. Male participants whose female partner is post-menopausal, and participants who are abstinent from heterosexual intercourse as part of their usual lifestyle will also be eligible.

   Male participants must agree to refrain from donating sperm from screening until study completion, including the follow up period, for at least 90 days after the last dose of study drug.
10. Provides written informed consent and is willing and able to undergo all study procedures and attend the scheduled follow up visit/s per protocol

Exclusion Criteria:

1. A positive reverse transcriptase polymerase chain reaction (RT-PCR) test or rapid antigen test (RAT), as applicable, for influenza A/B or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2; COVID-19) at screening or at time of admission to the CRU.

   Note: A nose and/or throat swab or saliva sample may be collected and analysed for COVID-19 at screening, and at one or multiple timepoints during the study as per local, state and national guidelines and per the standard practice at the CRU.
2. A history of Hepatitis B, Hepatitis C or human immunodeficiency virus (HIV) infection and/or a positive pre-study HIV, Hepatitis B surface antigen (HbsAg), total Hepatitis B core antibody (HBcAb), or positive Hepatitis C virus (HCV) antibody result within 3 months of screening
3. Impaired hepatic function as indicated by screening aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than or equal to 2 or total bilirubin greater than or equal to 1.5 x upper limit of normal (ULN), which remains above these limits if retested (i.e., due to a slightly elevated initial result or abnormalities in synthetic liver function tests that are judged by the Investigator to be clinically significant)
4. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of known Gilbert's syndrome or asymptomatic gallstones).
5. Any other serious medical condition or abnormality that, in the Investigator's judgement, precludes the participant's safe participation in and completion of the study.
6. A positive pre-study drug or alcohol screen. A positive drug or alcohol screen test result may be verified by re-testing (up to 1 false positive result permitted) and may be followed up at the discretion of the Investigator.
7. History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units for males or greater than 14 units for females. One unit is equivalent to 10 g of alcohol and the following can be used as a guide: a half-pint (~240 ml) of beer, 1 glass (125 mL) of wine or 1 (30 mL) measure of spirits.
8. The participant is unwilling to abstain from alcohol consumption from 24 hours prior to dosing until discharge from the CRU, and for 24 hours prior to all other outpatient visits to the CRU.
9. The participant is unwilling to abstain from smoking while domiciled at the CRU.
10. Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human or humanised antibodies, fusion proteins, ALT-100 excipients, or a history of drug or other allergy including severe allergic reaction that in the opinion of the Investigator, local MM or Sponsor medical representative, contraindicates their participation.
11. Participants receiving more than 2 weeks' treatment with immunosuppressive agents, excluding topical steroids, in the previous 3 months.
12. Participation in a clinical trial within 30 days before randomisation; use of any experimental therapy within 30 days or 5 half-lives prior to randomisation, whichever is greater; or use of any biologic therapy within 12 weeks or 5 half-lives prior to randomisation, whichever is greater.
13. Participants having received any type of vaccination within 2 weeks of the anticipated dosing event or are expected to be vaccinated within 2 weeks post-dosing.
14. Use of prescription or non-prescription drugs (except simple analgesics and topical steroids), including vitamins, herbal and dietary supplements (including St John's Wort) within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose of study drug, unless in the opinion of the Investigator, local MM and Sponsor medical representative the medication will not interfere with the study procedures or compromise participant safety.
15. Pregnant or breastfeeding WOCBP
16. Donation within the last 3 months of whole blood (greater than 499 mL) and/ or within 2 weeks of plasma.
17. Participant unable to provide written informed consent.
18. Unwilling or unable to follow protocol requirements, including attendance at follow up visit/s.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed by the incidence, frequency and dose-relationship of all adverse events | up to 120 days post ALT-100 infusion

SECONDARY OUTCOMES:
Plasma PK Parameter: Area under concentration-time curve from time 0 (pre-dose) to the last quantifiable data point (AUC0-t) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Plasma PK Parameter: Area under concentration-time curve from time 0 (pre-dose) extrapolated to infinity point (AUC0-infinity) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Plasma PK Parameter:: Maximum measured drug concentration (Cmax) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Plasma PK Parameter: Dose normalised Cmax (determined by Cmax/dose [D]) and dose normalised AUC determined by AUC/D) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Plasma PK Parameter: The percent of the AUC from time 0 (pre-dose) extrapolated to infinity determined by AUC/D) (%AUCextrap) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Plasma PK Parameter: Time of maximum concentration (Tmax) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Plasma PK Parameter: Terminal elimination rate constant (kel) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Plasma PK Parameter: Elimination half-life (T½) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Plasma PK Parameter: Total body clearance (CL) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Plasma PK Parameter: Volume of distribution at the terminal phase (Vz) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Plasma PK Parameter: Dose normalised Cmax (determined by Cmax/dose [D]) and dose normalised AUC (determined by AUC/D) | at 10, 20, 30, 45 minutes, and 1, 2, 4, 8, hours post start of ALT-100 infusion and on Days 2, 3, 8. 15, 22, 29, 60, 90 and 120.
Serum Immunogenicity: To investigate the presence of antibodies that bind to ALT-100, and if detected, to initiate characterisation of these anti-ALT-100 antibodies (anti-drug antibodies; ADA). | Presence of ADA in serum on Days 8, 15, 29, 60, 90 and 120 days following ALT-100 treatment

OTHER OUTCOMES:
Changes from baseline in cellular response with ALT-100 compared to placebo, as assessed by peripheral circulating neutrophil counts in whole blood | at 6, 24, and 48 hours, and 7, 14 and 28 days following ALT-100 treatment
Changes from baseline in cellular response with ALT-100 compared to placebo, as assessed by peripheral circulating monocyte counts in whole blood | at 6, 24, and 48 hours, and 7, 14 and 28 days following ALT-100 treatment
Changes from baseline in cellular response with ALT-100 compared to placebo, as assessed by peripheral circulating lymphocyte counts in whole blood | at 6, 24, and 48 hours, and 7, 14 and 28 days following ALT-100 treatment
Changes from baseline in plasma levels of extracellular nicotinamide phosphoribosyltransferase (eNAMPT) compared to the placebo control | at 6, 24, and 48 hours, and 7, 14 and 28 days following ALT-100 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joe GN Garcia, MD, Study Director — Aqualung Therapeutics; Thomas M Polasek, MBBS, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No